CLINICAL TRIAL: NCT04991077
Title: Interrupters of VAscular daMAge in Malignant Hypertension: Role of Inflammasome, Angiogenic and Vasoactive System
Brief Title: Interrupters of VAscular daMAge in Malignant Hypertension
Acronym: IVAMA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Other Study IDs: CHPAU2021/02
Record Dates: First submitted 2021-06-16; First posted 2021-08-05 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Malignant Hypertension
Keywords: malignant hypertension; severe hypertension; hypertensive emergency; pathophysiology; angiogenic system; inflammasome
MeSH Terms: conditions — Hypertension, Malignant; Hypertension; Hypertensive Crisis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients group: patients with malignant hypertension
  Interventions: Biological: analyse of angiogenic, vasoactive and VEGF systems
- Control group: patients with severe hypertension (Grade 2 or 3 hypertension)
  Interventions: Biological: analyse of angiogenic, vasoactive and VEGF systems

INTERVENTIONS:
Biological: analyse of angiogenic, vasoactive and VEGF systems — the angiogenic, vasoactive and VEGF systems will be analysed through blood and urine sampling. These samples will be collected at the time of malignant hypertension diagnosis and repeated one month later, in 30 patients (patients group). The same tests will be performed once in 15 patients with severe non-malignant hypertension, constituting the control group.

SUMMARY:
The pathophysiology of malignant hypertension is poorly understood. The objective of this translational research project is to evaluate the relationship between activation of vasoactive systems (renin-angiotensin and endothelin systems), angiogenic signal deficiency (VEGF and sFlt-1) and the occurrence of malignant hypertension episodes in humans.

DETAILED DESCRIPTION:
The pathophysiology of malignant hypertension is poorly understood. The current dogma is based on an overwhelming renin-angiotensin-aldosterone system activation, leading to arterial hypertension that overcomes target organ auto-regulatory mechanisms and leads to subacute microvascular lesions. However, some patients present with normal or lowered renin in the acute phase of malignant hypertension, suggesting other pathophysiological pathways. Malignant hypertension was reported following anti-VEGF treatment, suggesting that this pathway may be involved. Recent unpublished animal data highlight 1/ the possibility of severe deregulation of the VEGF (vascular endothelial growth factor) system in malignant hypertension 2/ the possibility of compensation of the vasculotoxic effects of VEGF deficiency by inflammasome components. These systems have never been studied together in human hypertension.

Investigators will analyze the angiogenic, vasoactive and VEGF systems through blood and urine sampling. These samples will be collected at the time of malignant hypertension diagnosis and repeated one month later in 30 patients. The same tests will be performed in 15 patients with severe non-malignant hypertension, constituting the control group.

ELIGIBILITY:
Inclusion Criteria:

Patients group :

* Patients included in the HAMA cohort
* Who is willing to take part in the IVAMA project

Control group :

* Grade 2 or 3 hypertension with office blood pressure measurement (above 160 and/or 100 mmHg for systolic and diastolic)
* Persistence of blood pressure above 160 / 100 mmHg on the average of 3 "attended" blood pressure measurements

Exclusion criteria:

Patients group :

* Age < 18 years old
* Patients with chronic renal failure of stage 3 or higher.
* Patients with any type of diabetes
* Patient in per partum
* Patients who cannot freely give their consent, or patients who refuse to participate
* Chronic dialysis patient

Control group:

* Evidence of subacute involvement of one of the following target organs: brain, kidney, eye, heart, thrombotic microangiopathy. Target organ impairment is defined in the inclusion criteria for the "Patients" group.
* Presence of known chronic kidney insufficiency of grade 3 or higher
* Chronic dialysis patient
* Diabetes of any type
* Patients who cannot freely give their consent, or patients who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient group: patient with malignant hypertension control group: paitent with severe hypertension
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
sFLT1 concentration at inclusion | at the end of study recrutment, an average of 11 month
  The primary endpoint will be the difference in sFLT1 concentrations between patients and controls at enrolment

SECONDARY OUTCOMES:
IL1ß concentration at inclusion | at the end of study recrutment, an average of 11 month
  Difference in IL1ß concentrations between patients and controls at enrolment
VEGF concentration at inclusion | at the end of study recrutment, an average of 11 month
  Difference in VEGF concentrations between patients and controls at enrolment
renin concentration at inclusion | at the end of study recrutment, an average of 11 month
  Difference in renin concentrations between patients and controls at enrolmentD30, and compare this evolution.
angiotensin concentration at inclusion | at the end of study recrutment, an average of 11 month
  Difference in angiotensin concentrations between patients and controls at enrolmentD30, and compare this evolution.
evolution of IL1ß concentration | through study completion, an average of 12 month
  Evaluation of the evolution of IL1ß concentration in the two groups between D0 and D30, and compare this evolution.
evolution of VEGF concentration | through study completion, an average of 12 month
  Evaluation of the evolution of VEGF concentration in the two groups between D0 and D30, and compare this evolution.
evolution of renin concentration | through study completion, an average of 12 month
  Evaluation of the evolution of renin concentration in the two groups between D0 and D30, and compare this evolution.
evolution of angiotensin concentration | through study completion, an average of 12 month
  Evaluation of the evolution of angiotensin concentration in the two groups between D0 and D30, and compare this evolution.
mutations in the genes of interest | through study completion, an average of 11 month
  comparison in the 2 groups of the frequency of mutations in the genes of interest underlying the vasoactive, angiogenic and VEGF systems

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Hôpital Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - Hôpital Bichat, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Chu Rangueil, Toulouse
  - CHU de Tours, Tours